CLINICAL TRIAL: NCT03843489
Title: SpO2 Accuracy In Vivo Testing for Neonates & Infants - Convenience Arterial Samples Compared to CO-Oximetry
Brief Title: SpO2 Accuracy In Vivo Testing for Neonates & Infants
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision
Sponsor: Medline Industries (Industry)
Collaborators: Clinimark, LLC (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PR2018-296
Record Dates: First submitted 2019-02-12; First posted 2019-02-18 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Pulse Oximetry

STUDY DESIGN:
Intervention Model Description: Hospital staff will place the pulse oximeter sensor(s) on one or both hand or feet of the neonate/infant and start the pulse oximeter data collection computer to record continuously. Each time an arterial CO-Oximeter sample is collected the data collection file will be marked by pressing the file marker key on the data collection computer. Information from each arterial CO-Oximeter sample will be written on the CRF. The arterial sample will always be measured in the reference co-oximeter. The sample may also be measured in the currently used AVOX 1000E.
  This study will only use arterial blood samples that are taken in the normal course of care; the sample size of the blood draw will not be altered for this study (sample size will not be increased from the normal course of care for any portion of this study).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- MEDLINE RENEWAL PULSE OXIMETRY SENSORS (Experimental): Reference sensors from the reprocessed oximeter device will be placed on each subject to evaluate the SpO2 accuracy and performance.
  Interventions: Device: MEDLINE RENEWAL PULSE OXIMETRY SENSORS
- Reference CO-oximetry sensor (Sham Comparator): A whole blood analyzer (CO-Oximeter) is used as the reference standard device for obtaining the functional SaO2 value from arterial blood samples obtained during the study.
  Interventions: Device: Reference CO-oximetry sensor

INTERVENTIONS:
Device: MEDLINE RENEWAL PULSE OXIMETRY SENSORS — An oximeter is a device used to transmit radiation at a known wavelength(s) through blood and to measure the blood oxygen saturation based on the amount of reflected or scattered radiation. Pulse oximetry monitoring is considered a standard physiological measurement and is used by clinicians in everyday situations to estimate arterial oxygen saturation. Because an arterial sample of blood is not required to make the measurement, the pulse oximeter can provide non-invasive real time information.
  Arms: MEDLINE RENEWAL PULSE OXIMETRY SENSORS
Device: Reference CO-oximetry sensor — A whole blood analyzer (CO-Oximeter) is used as the reference standard device for obtaining the functional SaO2 value from arterial blood samples obtained during the study.
  Arms: Reference CO-oximetry sensor

SUMMARY:
The purpose of this clinical study is to validate the oxygen saturation (SpO2) accuracy of various pulse oximetry systems and sensors (new designs and/or reprocessed) during non-motion conditions as compared to arterial blood samples, drawn in the normal course of patient care, assessed by CO-Oximetry in neonates and infants. The primary end goal is to provide supporting documentation for the SpO2 accuracy of these pulse oximetry systems. The secondary end goal is to provide data for evaluation of clinical impact of measured to calculated SaO2 and related issues.

DETAILED DESCRIPTION:
FDA Guidance for pulse oximeters (March 4, 2013), section 4.1.2, In vivo testing for SpO2 accuracy for neonates, calls for the devices to be first tested in adults during hypoxia tests with arterial samples compared to measured oxygen saturation. This has been previously completed on the devices that will be tested in this protocol. In order to verify safe clinical performance in the neonate, the FDA then requires testing using neonatal arterial samples that are collected in the normal course of care; which is the primary purpose of this protocol. As a secondary purpose the data will be utilized to evaluate the impact of calculated oxygen saturation versus measured oxygen saturation and related issues.

Neonates/infants who will have an arterial line or sheath placed in the normal course of care will be included in this study. The pulse oximeter sensor must be placed on the Neonates/infant's foot or hand. Neonates who either have repaired PDA but are having the placement of the sensor on the foot (which will be arterial blood only) will be allowed as long as other inclusion/exclusion criteria are met.

ELIGIBILITY:
Inclusion Criteria:

* Neonates/Infants up to 28 days old
* Neonates/Infants less than 5kg.

And one of the following:

Without PDA With a PDA with R-L shunting that will be repaired before arterial samples are taken

Exclusion Criteria:

* Physical malformation of feet or toes or other sensor sites which would limit the ability to place the sensors for the study.
* Neonates/Infants older than 28 days old.
* Neonates/Infants outside the weight range for the sensor (Greater than 5kg.)
* Neonates/Infants with unrepaired PDA. with PDA with R-L shunting
* Subjects who are undergoing bilirubin light therapy while samples are being obtained.

Max Age: 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-03-19 (Estimated); Primary Completion 2021-09-20 (Estimated); Study Completion 2021-09-20 (Estimated)

PRIMARY OUTCOMES:
Validation of SpO2 accuracy of pulse oximetry sensors | 4 hours
  To validate SpO2 accuracy performance of Sponsor sensors by an Accuracy Root Mean Square (Arms) value. Reference CO-Oximetry will be used as the basis for comparison for the investigational device SpO2 readings.

SECONDARY OUTCOMES:
Calculated oxygen saturation versus measured oxygen saturation | 4 hours
  The arterial sample will always be measured in the reference co-oximeter. The sample may also be measured in the currently used AVOX 1000E.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Deterding, MD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided